CLINICAL TRIAL: NCT04127812
Title: Evaluating a Mindful Eating Curriculum, "Savor the Flavor" to Promote Healthy Eating Among Head Start Preschool Children
Brief Title: Evaluating a Mindful Eating Curriculum, "Savor the Flavor"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Associate Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013064
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Eating Behavior
Keywords: mindfullness; eating; snacking; obesity; children
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Selected classrooms will receive the Savor the Flavor intervention. Data will be collected prior to and after the intervention. Children, their parent/guardian, and classroom teachers will participate in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savor the Flavor (Experimental): The "Savor the Flavor" curriculum is a series of five interactive lessons designed to teach children how to savor foods and slow down while eating by focusing on the sensory experience of eating. The intervention also teaches attention control techniques so that children are better able to delay consumption of high energy, low nutrition foods, when appropriate, as well as general mindfulness practices (e.g. breathing exercises). Lessons are delivered in the Head Start classroom by a nutrition educator.
  Interventions: Behavioral: Savor the Flavor

INTERVENTIONS:
Behavioral: Savor the Flavor — A series of five interactive classroom lessons focused on mindfulness in eating.

SUMMARY:
The overall goal of this study is to conduct a preliminary evaluation of the feasibility and efficacy of the "Savor the Flavor" intervention.

DETAILED DESCRIPTION:
The overall goal of this study is to conduct a preliminary evaluation of the feasibility and efficacy of the "Savor the Flavor" intervention. The goal of this curriculum is to teach children how to savor foods and slow down while eating by focusing on the sensory experience of eating. The intervention will also teach children attention control techniques so that they are better able to delay consumption of high energy, low nutrition foods, when appropriate.The study will also evaluate a modified version of the Eating in the Absence of Hunger task for use in a preschool classroom setting.

ELIGIBILITY:
Child Inclusion Criteria:

* Child must be enrolled in a Head Start preschool center
* Child must be between the ages of 2 and 6 years old

Child Exclusion Criteria:

* Food allergy or restriction to foods included in protocol

Parent Inclusion Criteria:

* Parent or other primary caregiver of a child enrolled in the study
* 18 years of age or older
* English speaking

Parent Exclusion Criteria:

- None

Teacher Inclusion Criteria:

* Actively employed as an early childhood education provider in the Head Start classroom where intervention is delivered
* 18 years of age or older

Teacher Exclusion Criteria:

- None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in eating in the absence of hunger from pre to post intervention | Pre intervention and at conclusion of 5 week intervention
  Children will be given seven minutes of free access to a variety of palatable snacks and toys during a time when they are not hungry (e.g. after a meal). Intake of snacks is determined by pre and post weighing the foods.

SECONDARY OUTCOMES:
Recall of Savor the Flavor steps | At conclusion of 5 week intervention
  Children will be asked to recall the five steps of "Savor the Flavor"
Acceptability of intervention | At conclusion of 5 week intervention
  Teachers will complete a questionnaire with scaled and open-ended questions about the feasibility and acceptability of the intervention

OTHER OUTCOMES:
Child body mass index | Measured once at any time between enrollment and conclusion of 5 week intervention
  Child height and weight will be measured and used to calculate body mass index (BMI). Age and sex specific BMI percentiles/z-scores will be calculated using CDC growth standards
Child Eating Behavior Questionnaire | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the Child Eating Behavior Questionnaire as part of a survey packet
Structure and Control in Parent Feeding | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the Structure and Control in Parent Feeding as part of a survey packet
USDA Food Security questionnaire | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the USDA food security questionnaire as part of a survey packet
External Food Responsiveness scale | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the External Food Responsiveness Scale as part of a survey packet
Eating in the Absence of Hunger scale | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the Eating in the Absence of Hunger Scale as part of a survey packet

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Savage, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available from the principal investigator upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication of primary outcomes.
Access Criteria: Access requests will be evaluated and approved at the principal investigator's discretion.